CLINICAL TRIAL: NCT00349323
Title: Community-Directed Treatment in the Control of Soil-Transmitted Helminths Among Children Aged 12-59 Months in Mazabuka District of Zambia
Brief Title: Community Directed Treatment of Soil-Transmitted Helminths Among Young Children in Zambia
Status: Completed | Type: Observational
Sponsor: DBL -Institute for Health Research and Development (Other)
Collaborators: Department of Community Medicine & Department of Biological Sciences (Unknown); University of Zambia (Other)
Other Study IDs: 2006-7041-83/hah
Record Dates: First submitted 2006-07-06; First posted 2006-07-07 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2008-02

CONDITIONS: Soil-Transmitted Helminth Infection; Growth
Keywords: Community directed treatment,; soil-transmitted helminth infections,; treatment coverage,; Zambia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Community directed treatment

SUMMARY:
The WHO Special Programme for Research and Training in Tropical Diseases (TDR) developed a Community-Directed Treatment (COMDT) approach, which has been adopted in the control of onchocerciasis and lymphatic filariasis. WHO has recommended the use of COMDT approach in the control of schistosomiasis and STH infections. The COMDT approach has been compared with the school based programmes in certain African countries,but not with the health-facility based approach.

The project will be implemented in Mazabuka district of Zambia where COMDT approach will be implemented in the catchment area of Rural Health Centres (RHC) as a supplement to the health-facility-based approach. After each round of treatmenttreatment coverage and factors responsible for the treatment coverage will be measured in both areas. The health impact of the health facility based approach with and without the COMDT approach will be compared. The effect of the COMDT as a control approach of STH infections will be monitored on infections in the community of children aged 12 to 59 months.

DETAILED DESCRIPTION:
Soil-transmitted helminth (STH) infections are of public health importance and widespread in large part of the world, particularly in the poorest sections of the populations residing in the least developed countries. The infections can be controlled by several measures, but currently delivering anthelminthic drugs through schools and health centres is believed to be the most effective as it takes advantage of existing infrastructure. In Zambia, anthelminthic drugs are delivered to children aged 12 to 59 months twice a year through health facilities during the child health promotion week. However, it has been observed that treatment coverage is low in certain areas. Therefore, there is a need to identify the factors associated with the treatment coverage patterns, and to provide evidence of an effective intervention approach that could increase the proportion of children receiving treatment.

The WHO Special Programme for Research and Training in Tropical Diseases (TDR) developed a Community-Directed Treatment (COMDT) approach, which has been adopted in the control of onchocerciasis and lymphatic filariasis. WHO has recommended the use of COMDT approach in the control of schistosomiasis and STH infections. The COMDT approach has been compared with the school based programmes in certain African countries, but has never been used in Zambia and never been compared with the health-facility based approach in the control of these infections in children below school age. It is against this background that this project is being proposed.

The project will be implemented in Mazabuka district of Zambia. Two Rural Health Centres (RHCs) will be selected in the district and mapped for treatment coverage of the health-facility based approach. Focus group discussions (FGDs) and in-depth interviews will be conducted with community members to explore the reasons for existing treatment coverage of the health facility approach. The COMDT approach will then be implemented in the catchment area of one of the RHCs as a supplement to the health-facility-based approach. After each round of treatment, coverage and factors influencing coverage will be measured in both areas. The health impact of the health facility based approach with and without the COMDT approach will be compared. Parameters for health impact will be child growth, prevalence and intensity of STH infections and number of illness episodes requiring treatment. The effect of the COMDT as a control approach of STH infections will be monitored on infections in the community of children aged 12 to 59 months, and the appropriateness of the approach will be evaluated using the African Programme for Onchocerciasis Control grading system. The whole project is expected to take 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-59 months

Exclusion Criteria:

* Severely ill children

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2006-08; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hikabasa Halwindi, M.phil, Principal Investigator — Department of Community Medicine, University of Zambia
Locations (1):
- Mazabuka District, Mazabuka, Zambia

REFERENCES:
- [Derived] Halwindi H, Magnussen P, Meyrowitsch D, Handema R, Siziya S, Olsen A. Effect on treatment coverage of adding community-directed treatment to the health facility-based approach of delivering anthelminthic drugs to under-five children during child health week in Mazabuka District, Zambia. Int Health. 2010 Dec;2(4):253-61. doi: 10.1016/j.inhe.2010.09.003. PMID 24037866